CLINICAL TRIAL: NCT01921972
Title: Competence Network - Dementia (BMBF) "Pharmacological and Psychosocial Treatment" (Modul E.2) Part II: The Efficacy of a Combination Regimen in Patients With Mild to Moderate Probable Alzheimer's Disease
Brief Title: The Efficacy of a Combination Regimen in Patients With Mild to Moderate Probable Alzheimer's Disease
Acronym: AD-Combi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Isabella Heuser, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Modul E.2 II
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Alzheimer's Disease
Keywords: AD, Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine and Placebo (Active Comparator): Subjects in this group will receive 4 weeks of 8 mg/day galantamine CR, followed by 4 weeks of 16 mg/day and from week 9 up to the end of the trial of 24 mg/day.
  Interventions: Drug: Galantamine CR; Drug: Placebo
- Galantamine and Memantine (Experimental): Galantamine titration will be performed as described above. Memantine titration will be performed over 4 weeks in steps of 5 mg/day up to 20mg/day (10 mg b.i.d.). 50 % of this group will receive galantamine first, 50 % of the group will receive memantine first to allow for differential qualitative evaluation of tolerability of a combination therapy.
  Interventions: Drug: Galantamine CR; Drug: Memantine

INTERVENTIONS:
Drug: Galantamine CR — 24 mg/day with dose-titration over twelve weeks
Drug: Memantine — memantine 10 mg b.i.d. with a dose titration of sixteen weeks
  Arms: Galantamine and Memantine
Drug: Placebo — Placebo will be similar in appearance to Memantine
  Arms: Galantamine and Placebo

SUMMARY:
This is a national multicenter, double-blind, randomized, parallel-group trial of 12 months in duration. Following a 4 week wash-out period, subjects will be randomized to one of 2 treatment groups: (1) galantamine CR 24 mg/day with dose-titration over twelve weeks[maintenance phase from week 9], (2) a combination of galantamine CR 24 mg/day plus memantine 10 mg b.i.d. with a dose titration of sixteen weeks (12 weeks for galantamine [maintenance phase from week 9], additional 4 weeks for memantine).

DETAILED DESCRIPTION:
Based on 1. the established efficacy of both, galantamine and memantine in subjects with Alzheimer's disease, 2. galantamine's dual mode of action being a cholinesterase inhibitor and an allosteric modulator of the nicotinic acetylcholine receptor (nAChR) an effect which might lead to enhanced neurotransmission in other neuronal populations, i.e., glutamatergic and GABAergic, 3. memantine's neuroprotective properties, which have been demonstrated in several experimental system, but not yet in a clinical setting the primary hypothesis is formulated that treatment with a combination of galantamine plus memantine, which may exert additional effects on the level of neurotransmitter modulation, will reduce the memory/cognitive problems in AD patients. The effects of the combination therapy will be compared to galantamine effects alone.

As a secondary hypothesis, it is proposed that a combination treatment with galantamine plus memantine could conceivably slow disease progression and/or delay the progression of dementia in probable AD. It is reasonable to assume that the effect will be clearer with a combination therapy (galantamine, memantine) than with cholinesterase inhibitors alone which have been evaluated in long-term clinical trials (rivastigmine, donepezil, galantamine). To corroborate a potential disease modifying effect and to more reliably separate it from a purely symptomatic effect, the disease progress will not only be tracked by clinical measures (CDR rating), but also by using volumetric MRI techniques. Fox et al. have developed a sensitive method to follow changes in overall brain volume over time. In 'normal' ageing about 0.2%/year (SD 0.3%) change in brain volume is documented, whereas in AD, changes of 2.8%/year (SD 1%) are measured. People 'at risk' for developing AD show changes of about 1.5%/year. Recently it was established that rates of hippocampal atrophy correlate with change in clinical status in ageing ('conversion') and AD. Overall, brain atrophy or MRI delineated hippocampal volumes and memory decline seem to be clearly linked. The project will prospectively investigate the validity of investigations of hippocampal volume in assessing therapeutic effects in AD. MR-proton-spectroscopy provides consistent evidence that the neuronal marker Nacetylaspartat (NAA) is reduced in AD, whereas the role of myo-inositol, choline and creatine is less clear. NAA is thought to be present exclusively in neurons in gray matter and in their axonal processes in white matter and not in glial cells. NAA signal loss suggests neuronal loss when it is observed in gray matter and loss of or damage to axonal structures when it is observed in white matter. A correlation of NAA decrease in tissue samples of patients with AD with the number of senile plaques and neurofibrillary tangles was reported. Recent results indicate that the severity of dementia in patients with AD is positively correlated with the decrease in NAA/Cr only in the parietal cortex and in the temporal lobe. These data are consistent with the observation that the amount of synaptic loss is the dominant indicator of dementia in AD. The cognitive decline in patients with AD may be linked with a neuronal loss or dysfunction preferentially in the temporoparietal association cortex. This project will prospectively investigate the validity of spectroscopic abnormalities in assessing therapeutic effects in AD.

The primary objective of this trial is to establish the hypothesis that a combination of galantamine plus memantine improves memory/cognitive performance to a larger extent than galantamine monotherapy in AD subjects after one year of double-blind treatment.

Memory/cognitive performance will be assessed with the ADAS-cog/11. The confirmatory statistical assessment of this hypothesis will be based on the change of the ADAS-cog/11 from baseline to the end of the treatment period.

Additional endpoint variables to be assessed in an exploratory manner in parallel to the ADAS-cog are:

* Preservation of functionality as assessed using the ADCS-ADL/AD scale.
* Global rating of dementia as assessed using the CDR rating instrument.
* Neuropsychiatric symptoms as assessed using the NPI rating instrument.
* Resource utilization as assessed using the RUD rating instrument.
* Caregiver burden as assessed using the burden interview (BI).
* Safety with adverse event reports, laboratory parameters, vital signs, physical examination and ECG

The secondary hypothesis states that the combination therapy with galantamine plus memantine is more effective than galantamine alone in delaying clinical progression of dementia in this population over an observation period of one year. Global severity of dementia will be assessed with the CDR scale.

Supplementary endpoint criteria for this hypothesis are:

* Reduction in the rate of serial MRI determined brain (hippocampal) atrophy and of MRS-based parameters.
* Safety with adverse event reports, laboratory parameters, vital signs, physical examination and ECG.

Further analyses of sub-groups (e.g., determined by biological variables) or biological outcome measures investigated by the diagnostic module with respect to the above measures are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate, as indicated by written informed consent of the patient. The competence of the participating patient has to be assessed by a physician who is not involved in this trial.
2. Male or postmenopausal female outpatients.
3. Age of > 50 years at time of randomization.
4. Diagnosis of probable Alzheimer's Disease (according to NINCDS-ADRDA criteria).
5. Clinical and psychometric rating cut-off score (valid at randomisation): MMSE range of 15 to 26 points.
6. MRI brain scan not older than 12 months (before randomization) compatible with the diagnosis of Alzheimer's Disease. (The MRI brain scan must be repeated if older than 12 months or if clinically indicated).
7. Patient being ambulatory having adequate vision and hearing abilities to allow neuropsychological testing.
8. Patient with a knowledgeable, cooperative, reliable caregiver/informant who is willing to follow the study procedure as indicated by written informed consent.

Exclusion Criteria:

1. Dementia of any other type than AD:

   1. vascular dementia

      * HIS Score (modified acc. to Rosen) > 5 or
      * evidence for VD acc. to NINCDS-AIREN criteria.
   2. depressive pseudodementia defined acc. to DSM-IV criteria for major depression.
   3. other non-AD dementia.
2. Significant neurological disease other than AD, such as cerebral tumor, Huntington's disease, Parkinson's disease, normal pressure hydrocephalus, subdural hematoma, mental retardation, history of brain surgery or serious head trauma with residual deficits.
3. Diagnosis of psychosis (requiring hospitalization or antipsychotic therapy for more than two weeks) within the past 10 years not associated with AD or a diagnosis of alcoholism or drug dependence within the past 10 years.
4. History of epileptic seizures or patient receiving antiepileptic drugs.
5. Abnormal laboratory test results considered clinically relevant for dementia: e.g., electrolyte changes, folate deficiency, vitamin B12 deficiency, pathological thyroid function (T3 and TSH levels), positive syphilis serology.
6. Patient who, in the opinion of the investigator, is suffering from an acute or poorly controlled illness, such as:

   1. Presently uncontrolled hypertension (> 180 mmHg systolic or > 100 mmHg diastolic).
   2. Myocardial infarction within the last six months.
   3. Patient with uncompensated congestive heart failure (NYHA Class III or IV)
   4. Severe renal, hepatic or gastrointestinal disease, which could alter absorption, metabolism or excretion of the trial drug.
   5. Serum creatinine > 130 μmol/l or 1.5 mg/dl, transaminases (ALAT, ASAT) or GGT > twice the upper limit of normal range.
   6. Uncontrolled diabetes on entry into the double-blind phase of the research project (fasting blood glucose > 10.0 mmol/l or 180 mg/dl in repeated tests) or patient requiring insulin treatment.
7. Patient taking any inadmissible medication, such as:

   * Any investigational drug.
   * Anticonvulsants (incl. barbiturates).
   * Anti-Parkinson agents.
   * Dopaminergic agents.
   * Amantadine.
   * Antimuscarinic agents (i. e., anticholinergics).
   * Selegiline, MAOI.
8. Any condition that precludes cooperation with the tests or other investigations during the study (e.g., seeing or hearing loss, relevant confusion or agitation, musculoskeletal disorders, contraindication for magnetic resonance imaging, i.e., presence of pacemaker, metallic implants in high risk areas, presence of metallic material in high risk areas, history of claustrophobia. Hip implants are not contraindicated).
9. Patient has participated in an investigational clinical trial during the last 2 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2004-11; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
ADAScog/11 | change from Baseline to 12 months of treatment
  Alzheimer's Disease Assessment Scale (ADAS-cog/11) The ADAS consists of two parts - a cognitive subscale and a behavioral subscale. The behavioural subscale will not be used in this trial. The cognitive subscale, the ADAS-cog/11, consisting of Word Recall and Word Recognition memory tests, Object and Finger Naming, Commands, Constructional Praxis, Ideational Praxis, Orientation, Remembering Test Instructions, Spoken Language Ability, Comprehension of Spoken Language and Word Finding Difficulty will be the primary variable in this trial. In this trial the German version of the ADAS-cog/11 will be employed (Ihl & Weyer, 1993).

SECONDARY OUTCOMES:
ADCS-ADL | change from Baseline to 12 months of treatment
  The ability to perform activities of daily living will be assessed using the AD version of the Alzheimer's Disease Cooperative Study ADL inventory (Galasko et al., 1997, 2004). This instrument comprises questions about 23 basic and instrumental ADLs. For each ADL, the scores range from 0 (non-performance of the activity or the need for extensive help) to the highest score (representing independent performance of the activity). The total score ranges from 0 (no function) to 78 (maximal function).
Clinical Dementia Rating | change from Baseline to 12 months of treatment
  The CDR Scale is a clinician-rated dementia staging system that tracks the progression of cognitive and functional deterioration. Scores are on a scale of 0 - 5, with 0 = no dementia, 0.5 = questionable dementia, 1 = mild dementia, 2 = moderate dementia, 3 = severe dementia, 4 = profound dementia, and 5 = terminal dementia. Cognitive and functional abilities that are assessed are memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care. Memory is considered the primary driver for scoring with the other categories secondary.
Neuropsychiatric Inventory NPI | change from Baseline to 12 months of treatment
  The Neuropsychiatric Inventory (Cummings et al., 1994) is used to assess 10 areas of non-cognitive symptoms which are common in dementia, including delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, and aberrant motor activity. The NPI uses a screening strategy to minimize administration time. Interrater reliability and test-retest reliability are acceptable.
Resource Utilization of Dementia Scale (RUD) | change from Baseline to 12 months of treatment
  For each patient, use of medical and social services will be determined using the Resource Utilization of Dementia Scale (Wimo et al., 1998). This instrument is used to rate the primary caregiver (time spent on caring, occupational status, use of medical and social services, use of medications) and the patient (living arrangement, nursing home and hospital admissions, use of medical and social services) to estimate healthcare cost
Burden Interview (BI) | change from Baseline to 12 months of treatment
  The Burden Interview (Zarit & Zarit, 1983, 1990) has been designed to assess the stress experienced by family caregivers of elderly and disabled persons. It can be completed by caregivers themselves or as part of an interview. Caregivers are asked to respond to a series of 22 items about the impact of the patient's disabilities on their life. For each item caregivers are to indicate how often they have felt that way: never, rarely, sometimes, quite frequently, or nearly always.
  The Burden Interview is scored by summing the responses of the individual items. The total score ranges from 0 to 88. Higher scores indicate greater caregiver distress.
Adverse Event Reports | 12 months of treatment
Rate of brain atrophy | change from baseline to 12 months of treatment
  Serial volumetric MRI will generate data-sets used for whole brain rate of atrophy determinations, hippocampal rate of atrophy measurements as well as MR-spectroscopic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Heuser, Prof. Dr., Study Director — Free University of Berlin; Wolfgang Maier, Prof. Dr., Principal Investigator — University of Bonn; Wolfgang Gaebel, Prof. Dr., Principal Investigator — Heinrich-Heine University, Duesseldorf; Johannes Kornhuber, Prof. Dr., Principal Investigator — University of Erlangen-Nürnberg; Konrad Maurer, Prof. Dr., Principal Investigator — University of Frankfurt; C H Lücking, Prof. Dr., Principal Investigator — University of Freiburg; Eckhart Rüther, Prof. Dr., Principal Investigator — University of Göttingen; Mathias Berger, Prof. Dr., Principal Investigator — University of Freiburg; Dieter Naber, Prof. Dr., Principal Investigator — University of Hamburg-Eppendorf; Christoph Mundt, Prof. Dr., Principal Investigator — Heidelberg University; Lutz Frölich, Prof. Dr., Principal Investigator — Heidelberg University; Lutz Frölich, Prof. Dr., Study Director — Central Institute of Mental Health; Fritz A Henn, Prof. Dr., Principal Investigator — Central Institute of Mental Health; Matthias C Angermeyer, Prof. Dr., Principal Investigator — LMU München; Hans Förstl, Prof. Dr., Principal Investigator — Technical University of Munich; Peter Falkai, Prof. Dr., Principal Investigator — Universitäts-Nervenklinik Homburg

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] Peters O, Fuentes M, Joachim LK, Jessen F, Luckhaus C, Kornhuber J, Pantel J, Hull M, Schmidtke K, Ruther E, Moller HJ, Kurz A, Wiltfang J, Maier W, Wiese B, Frolich L, Heuser I. Combined treatment with memantine and galantamine-CR compared with galantamine-CR only in antidementia drug naive patients with mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2015 Oct 19;1(3):198-204. doi: 10.1016/j.trci.2015.10.001. eCollection 2015 Nov. PMID 29854939